CLINICAL TRIAL: NCT03430674
Title: Evaluation of an Exercise Intervention for Vincristine Induced Peripheral Neuropathy in Pediatric Cancer Patients
Acronym: Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jamie Renbarger, Professor of Pediatric Cancer Research, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1708708583
Record Dates: First submitted 2017-11-07; First posted 2018-02-13 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Clinic and at home exercise sessions.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise, questionnaires and blood draws.

SUMMARY:
The purpose of this study is to better understand whether or not children with ALL can complete an exercise program during treatment and whether or not that program may impact peripheral neuropathy. Researchers will also study changes in the blood and body that may occur during the program by collecting samples of blood at various times during the study.

Aim 1: Evaluate the feasibility and acceptability of EX as an intervention for VIPN in pediatric patients with ALL.

Aim 2: Estimate preliminary effect sizes of the EX intervention.

DETAILED DESCRIPTION:
Baseline visit (week 6):

This visit may take up to 1.5 hours total.

* The subject's exercise therapist will meet with them to discuss what they can expect throughout the program period. The subject will receive their exercise DVD to be used for at-home exercise sessions.
* The subject will be asked questions about how they are feeling and their general well-being. The subject will also be asked to complete several questionnaires about their neuropathy, confidence level about completing the program, support and expectations.
* The subject will be given a Fitbit with instructions about how and when to use it.
* The subject will have a sample of blood collected (15mL or about 1 tablespoon). The study team will time this blood draw to occur when they are already having blood drawn for routine clinical treatment.
* The subject will have a physical fitness test, which includes body measurements such as weight, height and blood pressure; also tests for physical strength, endurance and oxygen consumption. At the same time the subject is given the physical fitness test they will also be asked to not eat for 1 hour before this session.
* The subject will complete their first exercise session with their therapist.

Weeks 6-13:

During weeks 6-13 (8 weeks total), the subject will be asked to exercise for at least 15 minutes 6 times per week using the instructional DVD that was provided to them. The exercise the subject does will be tailored to their age range (either age 5-10 or 11-18) and will consist of strengthening and aerobic activities. The subject will also be asked to keep an exercise log that is provided by the study to record their exercise activity including how they felt when they exercised. The subject will be asked to perform one of their exercise sessions during weeks 8, 10, and 12 at Riley Hospital with their exercise therapist. The study team will coordinate this visit to occur during one of their regularly scheduled office visits. Post-program visit (week 14) This visit may take up to 1.5 hours total.

* The subject will be asked questions about how they are feeling and their general well-being. The subject will also be asked to complete several questionnaires about your neuropathy, confidence level about completing the program, support and expectations.
* The subject will have a sample of blood collected (15mL or about 1 tablespoon). The study team will time this blood draw to occur when they are already having blood drawn for routine clinical treatment.
* The subject will repeat the physical fitness test, which includes body measurements such as weight, height and blood pressure; also tests for physical strength, endurance and oxygen consumption. During the last session (week 14) the subject will also be asked to not eat for 1 hour before this session.
* The subject will be asked to complete a satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for this study if they are:

  1. age ≥ 5 and ≤ 18 years,
  2. have been diagnosed with acute lymphoblastic leukemia (ALL),
  3. will undergo the standard of care treatment for ALL with vincristine.
  4. will have a TNS-PV score of >3 at week 6

Exclusion Criteria:

* Participants will be ineligible for this study if they have:

  1. baseline peripheral neuropathy greater than grade 1 (prior to receiving any doses of vincristine),
  2. evidence of significant liver dysfunction,
  3. Down's Syndrome,
  4. pregnancy,
  5. severe illness or infection,
  6. current active treatment with erythropoietin,
  7. administration of vitamin supplements above 100% of the recommended daily allowance

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Renbarger, MD, Principal Investigator — Riley Hospital for Children - Indiana University
Locations (1):
- Riley Hospital for Children - Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Exercise Intervention: Interventions administered for clinic and at home exercise sessions: Exercise-15 minute sessions daily that include resistance and aerobic training. All training sessions will be provided via an online video they can access at any time. In addition, each session will address 3 core, 3 lower body and 3 upper body exercises that will last 50 seconds each for a total of 10 minutes.
Arm/Group | Exercise Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 16 [5 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline Neuropathy [Mean (Inter-Quartile Range); unit: units on a scale] — Total Neuropathy Score Pediatric Version; Range for each subscale is 0 to 4 with 0 being normal and 4 being the worst neuropathy. The total range is 0-36.
  units on a scale | 8 [4 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Greater Than 50% Compliance to Exercise Regimen
Description: Subjects will complete greater than 50% of exercise sessions during 8 week intervention. Subject report satisfaction with the intervention via questionnaires.
Time Frame: 8 weeks
Population: Looking at % sessions completed during 8 week program per subject.
Measure: Count of Participants; unit: Participants
Groups:
- Feasibility: 50 % compliance
Arm/Group | Feasibility
Number analyzed (Participants) | 10
Participants | 0

2. Primary Outcome: Acceptability - Parent Satisfaction Survey
Description: Parents will also be asked to complete a satisfaction survey regarding the exercise program, DVDs, and therapist support. The satisfaction survey consists of 13 items. Scores were on a Likert scale 1-5, 1 - strongly disagree and 5 - strongly agree. The total range is 13-65 with 65 being the greatest satisfaction possible and 13 being the worst satisfaction possible.
Time Frame: 8 weeks
Population: Any parent or caregiver with a child involved in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Intervention
Number analyzed (Participants) | 8
score on a scale | 4.096 (0.301)

3. Secondary Outcome: Acceptability - Patient Satisfaction Survey
Description: Patients will provide feedback on the exercise program, DVDs, and therapist support. The satisfaction survey consists of 13 items. The scale is 1-5 with 1 - strongly disagree and 5 - strongly agree. The total range is 13-65 with 65 being the greatest satisfaction possible and 13 being the worst satisfaction possible.
Time Frame: 8 weeks
Population: Patients over the age of 5. Scores were averaged from Likert scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Intervention
Number analyzed (Participants) | 7
score on a scale | 3.945 (0.365)

4. Secondary Outcome: Pediatric Neuropathy
Description: Total Neuropathy Score Pediatric Version; Range for each subscale is 0 to 4 with 0 being normal and 4 being the worst neuropathy. The total range is 0-36. 0 being no neuropathy. 36 being highest neuropathy possible.
Time Frame: 8 weeks
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- Post Intervention Neuropathy: Exercise Intervention Group
Arm/Group | Post Intervention Neuropathy
Number analyzed (Participants) | 10
score on a scale | 6 [5 to 7]

5. Secondary Outcome: Quality of Life - Changes in Quality of Life From Pre Intervention to Post Intervention a Total of 8 Weeks.
Description: Quality of Life: Pediatric Quality of Life Inventory; Each is 0 to 4 with 0 being never and 4 being almost always. The total scale score, the mean is computed as the sum of all the items over the number of items answered on all the scales. The difference between pre and post QOL scores. Total scale score consists of 4 dimensions, physical, emotional, social, and school functioning. Scores are transformed on a scale from 0-100. The greater the score the better the quality of life.
Time Frame: Baseline and 8 weeks
Population: The difference between pre and post intervention score is the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Post Intervention: Exercise Intervention Group
Arm/Group | Post Intervention
Number analyzed (Participants) | 6
score on a scale | 8.17 (14.81)

6. Secondary Outcome: PDGF-BB Levels (Platelet Derived Growth Factor)
Description: Changes in PDGF-BB (Platelet Derived Growth Factor) levels in plasma from pre to post intervention.
Time Frame: Baseline (T1=week 6) and T2=week 14
Measure: Mean (Standard Deviation); unit: percentage of baseline
Groups:
- Platelet Derived Growth Factor: Exercise Intervention Group Platelet Derived Growth Factor
Arm/Group | Platelet Derived Growth Factor
Number analyzed (Participants) | 10
percentage of baseline | 66.03 (186.21)

7. Secondary Outcome: NGF (Nerve Growth Factor)
Description: Change in NGF (Nerve Growth Factor) in plasma from pre to post intervention.
Time Frame: Baseline (T1=week 6) and T2=week 14
Measure: Mean (Standard Deviation); unit: percentage of baseline NGF
Groups:
- Nerve Growth Factor: Exercise Intervention Group
Arm/Group | Nerve Growth Factor
Number analyzed (Participants) | 10
percentage of baseline NGF | 37.98 (144.42)

8. Secondary Outcome: Quality of Life as a Result in Changes in Neuropathy Scores.
Description: Analyzing the correlation of changes in quality of life scores with neuropathy scores using Pearson's correlation coefficient.
Time Frame: 8 weeks
Population: Changes in neuropathy scores as correlated with quality of life scores.
Measure: Number; unit: Pearson's correlation coefficient
Arm/Group | Post Intervention Neuropathy
Number analyzed (Participants) | 4
Pearson's correlation coefficient | 0.80

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Exercise Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03430674/Prot_SAP_000.pdf